CLINICAL TRIAL: NCT01984736
Title: A Multi-Center, Open-Label Phase I Study to Investigate the Effect of Different Degrees of Hepatic Impairment on the Single-Dose Pharmacokinetics of EVP-6124 in Patients With Hepatic Impairment Compared to Subjects With Normal Hepatic Function
Brief Title: EVP-6124 Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVP-6124-020; 2012-004467-53 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-11-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Hepatic Impairment
Keywords: Pharmacokinetic; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EVP-6124, single dose (Experimental): Single dose, Tablet, single administration, Day 1
  Interventions: Drug: Experimental: EVP-6124

INTERVENTIONS:
Drug: Experimental: EVP-6124

SUMMARY:
The purpose of this study is to assess the pharmacokinetics of EVP-6124 and metabolites after a single oral dose in subjects with mild, moderate and severe hepatic impairment compared with subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects age 18 to 65 years (both inclusive).
* Able to understand and willing to sign the Informed Consent Form and able to comply with the study restrictions.
* Females may enroll if they are:

  1. documented to be surgically sterile or postmenopausal (amenorrhoea greater than 1 year and follicle stimulating hormone,FSH, greater than or equal to 30 mU/mL), or
  2. practicing true abstinence and having a negative urine pregnancy test at Screening and Day -1, or
  3. using double barrier contraception protection, out of which one should be a physical barrier method, such as adequate hormonal method (eg, contraceptive implants, injectables, oral contraceptives) and/or non-hormonal methods (eg, intrauterine device, condom, diaphragm or spermicides) from Screening or at least 2 weeks prior to study drug administration (whichever is earlier) until 30 days after intake of study medication and having a negative urine pregnancy test at Screening and Day -1.
* Males with partners of childbearing potential may be enrolled if they are:

  1. documented to be surgically sterile (vasectomy), or
  2. practicing true abstinence, or
  3. using adequate double barrier contraception method, out of which one should be a physical barrier for 90 days after the drug intake.
* BMI 18.0 - 35.0 kg/m2, inclusive, where BMI (kg/m2) = body weight (kg) / height2 (m2).
* Patients with diabetes mellitus can be included provided that the disease is controlled (as judged by the PI).

Exclusion Criteria:

* Clinically relevant abnormal history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at the pre-trial screening assessment that the Investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer except for conditions associated with hepatic impairment in subjects with liver cirrhosis (Groups 1 and 2).
* Surgery (eg stomach bypass) or medical condition that might significantly affect absorption of medicines (as judged by the PI).
* Uncontrolled treated/untreated hypertension (defined as a mean of 3 repeated measurements for systolic blood pressure greater than or equal to 160 mmHg and/or diastolic blood pressure greater than or equal to 105 mmHg); current or documented history of repeated clinically significant hypotension or severe episodes of orthostatic hypotension (systolic blood pressure <90 mmHg and/or diastolic blood pressure less than 50 mmHg).
* History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
* Participation in another investigational drug trial within 30 days prior to dosing (or 5 times the half-life of the drug, whichever is longer) or exposure to more than three new investigational agents within 12 months prior to enrolment.
* Acute illness within 14 days prior to dosing unless mild in severity and approved by the Investigator and Sponsor's medical representative.
* Presence of active infection requiring antibiotics.
* History of cancer (judged not to be in full remission) or presence of cancer (except basal cell skin cancer or squamous cell skin cancer) as judged by the Investigator.
* Positive urine drug screen (if not due to concomitant medication) or alcohol breath test at Screening and/or Day -1.
* History of drug abuse within the last 2 years.
* Ingestion of alcohol and caffeine within 24 hours prior to dosing and during confinement. Regular alcohol consumption must not exceed 21 units for males and 14 units for females per week (1 unit equals 340 mL of beer, 115 mL of wine or 43 mL of spirits).
* Smoking of more than 10 cigarettes or equivalent per day.
* Concomitant use of medications known to be strong cytochrome (CYP) P450 inducers or inhibitors within 21 days prior to study drug administration.
* Consumption of grapefruit, grapefruit juice, pomelo, or Seville oranges within 7 days prior to study drug administration and during the study conduct.
* Positive serology for anti-Human immunodeficiency virus subtype 1 or 2.
* Loss of more than 450 mL blood during the 3 months before the trial (eg, as a blood donor).
* Female subjects who are pregnant, nursing, or planning to become pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of EVP-6124 and metabolites after a single oral dose in subjects with mild, moderate and severe hepatic impairment compared with subjects with normal hepatic function. | Oral clearance of EVP-6124, Maximum plasma concentration, Terminal elimination half life, and Total area under the plasma concentration time curve from time t to time infinity [Time Frame 0-288 hours postdose]

SECONDARY OUTCOMES:
Safety and tolerability of oral EVP-6124 in subjects with mild, moderate and severe hepatic impairment and in subjects with normal hepatic function. | Day 1 to Day 13 or Early Termination
  Adverse events, serious adverse events, and concomitant medications will be continuously monitored starting after the time of informed consent through the safety follow-up visit. Assessments will be made via recording of adverse events, concomitant medications, laboratory safety tests, vital signs, 12-lead ECGs and physical examinations.

CONTACTS AND LOCATIONS:
Locations (3):
- Jankovcova 1569/2c, 17000 Praha 7, Czechia
- Ul. Seczkowa 20b/8, Warszawa, Mazowieckie, 02-793, Poland
- Bardosova 2/A 83101 Bratislava, Slovakia